CLINICAL TRIAL: NCT07388342
Title: Diagnostic Accuracy of ECG-less Gated Cardiac CT in Resuscitated Cardiac Arrest Survivors
Brief Title: Diagnostic Accuracy of ECG-less Gated Cardiac CT in Resuscitated Cardiac Arrest Survivors Without ST Elevation Myocardial Infarction
Acronym: OPEN CCTArrest
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Bert Popelier, Principle investigator, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1432025000122
Record Dates: First submitted 2025-10-15; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest (CA); Myocardial Infarction (MI)
Keywords: Cardiac Arrest; Myocardial Infarction; Coronary Computed Tomography Angiography (CCTA)
MeSH Terms: conditions — Heart Arrest; Myocardial Infarction

STUDY DESIGN:
Masking Description: The results of cardiac part of the CT scan will be masked for the clinician (as there is no sufficient validation of this technique in this specific clinical setting) and for the interventional cardiologist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cardiac arrest survivor without STEMI (Experimental): Survivor of a cardiac arrest without STEMI, meeting inclusion criteria and no exclusion criteria, with informed consent from either the patient or his/her representative.
  Interventions: Device: ECG-less gated cardiac CT

INTERVENTIONS:
Device: ECG-less gated cardiac CT — Perform ECG-less gated cardiac CT during the CT scan routinely executed after survival of cardiac arrest in patients without STEMI.

SUMMARY:
In a significant portion of patients surviving a cardiac arrest, the event is caused by a myocardial infarction (a narrowing or blockage of one or more blood vessels that supply blood to the heart, the coronary arteries). In some people, this is immediately evident from basic tests; in others, it is more difficult to predict with the currently available tests whether this (or something else) caused the cardiac arrest. We investigate a technique that allows us to also assess the coronary arteries on the CT scan that is performed in patients surviving a cardiac arrest. The coronary angiography is currently the best exam we have for examining the coronary arteries, but it has some disadvantages. Compared to the CT scan, it takes more time, needs a more complex access to the blood vessels, and has some rare but relevant possible complications. The major advantage of the coronary angiography is that there is the possibility of immediate treatment of a narrowed/blocked blood vessel of the heart. The current guidelines advice an urgent coronary angiography when a clear myocardial infarction is suggested on the electrocardiogram, but not when there is no clear indication of myocardial infarction. Nonetheless, a relevant portion (more or less 40%) of the patients without a clearly abnormal electrocardiogram, still have an important problem in the blood vessels of the heart. We aim to determine whether the CT scan provides accurate information about the condition of the blood vessels of the heart. The CT scan was already well examined for this purpose before, but in the currently conventional way it needs preparation with extra monitoring and administration of medication, which would lead to loss of precious time and potentially dangerous side effects of these drugs in this critical situation. For that reason, a new software modality was developed that allows us to examine the coronary arteries in the same CT scan, without need for additional monitoring or medication administration. It does not need additional contrast administration (the dye necessary for optimal evaluation of some diseases).

The goal of this study is to determine whether this new technique gives us the correct information about the coronary arteries. This means we acquire the images of the heart in the same scan, and verify the results with the conventional coronary angiography. If the technique provides accurate information, it could lead to a better selection of patients we need to urgently refer for a coronary angiography and to defer the exam in those who have normal coronary arteries on the scan.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is the most important treatable cause of cardiac arrest. In contrast with cardiac arrest survivors with ST elevation myocardial infarction (STEMI), current guidelines do not recommend unselected/routine urgent invasive coronary angiography (ICA) in the patients with cardiac arrest without STEMI. This recommendation reflects existing evidence indicating that immediate invasive strategies may not confer significant benefit in this population and may even be harmful, while another ongoing randomized controlled trial is investigating this. Nevertheless, in COACT, a landmark trial investigating a strategy of immediate versus delayed coronary angiography in out-of-hospital cardiac arrest patients without STEMI, one or more culprit coronary lesions responsible for triggering cardiac arrest were identified in 40% of the total patient population. The question remains pertinent whether well selected cardiac arrest survivors without STEMI can benefit from early ICA. Yet, current available clinical tools fail to identify these patients. Markers such as clinical history, echocardiographic abnormalities, arrest rhythm (shockable/non-shockable), ECG changes other than ST-segment elevation and troponin levels lack sufficient sensitivity and specificity in a cardiac arrest setting for predicting ACS requiring intervention.

The diagnostic value of ECG-gated cardiac computed tomography angiography (CCTA) for detection of both acute and chronic coronary artery syndrome is well established, with recent evidence demonstrating the additional value of fractional flow reserve (FFR)-CT in ACS. Nonetheless, the need for ECG-gating remains a limitation.

Recently an ECG-less CCTA modality was developed, but its diagnostic accuracy is still under validation. ECG-less cardiac or coronary CT angiography (CCTA) allows cardiac imaging without requiring an ECG signal from the patient. Thus, it eliminates the steps associated with using a patient-attached ECG monitor: skin preparation, attaching the ECG leads, checking impedance, and confirming that the leads provide an adequate ECG signal to the scanning system. Therefore, workflow is optimized, which is critical in an emergency setting. In situations where it is difficult to attach the ECG leads, such as patients in a resuscitation setting who already have diagnostic ECG leads in place or other instrumentation, it is also advantageous that there is no need for an ECG signal.

Cardiac arrest patients without STEMI and with no evident non-cardiac cause generally undergo CT imaging of head and chest for evaluation of potential causes of cardiac arrest (e.g. pulmonary embolism, acute aortic dissection, intracranial hemorrhage). While ECG-gated CCTA is considered the optimal modality for non-invasive coronary imaging, ECG-less CCTA might offer a highly interesting alternative with the advantages mentioned earlier. Other benefits include no substantially longer scanning time, no need for additional contrast injection or administration of betablockers.

ECG-less Cardiac software is an FDA-approved cardiac scan mode that essentially utilizes existing CT system scan technology. The system uses a wide detector coverage of 160mm to provide full heart coverage and a fast gantry speed of 0.23 seconds per rotation to perform imaging in a single cardiac cycle. An estimate of the heart rhythm has to be provided, which is often readily available because emergency patients are already monitored. Based on the heart rhythm the scanner simulates an ECG signal. This simulated ECG signal provides virtual gating of the scan. The acquisition can be performed during a full heart cycle or three-quarters or half cycle, depending on how fast the heart rhythm is. The existing cardiac software options of SmartPhase (automated phase selection) and SnapShot Freeze 2 (optimized volume registration) amplify the quality of the images and correct for motion.

Patients are scanned using a Revolution Apex Elite system (GE Healthcare, Waukesha, WI -USA). The investigators use a hyperdrive pulmonary CT angiography (523mm/s with 0.28s/rotation gantry speed). After a short delay of a few seconds (5-12 sec), allowing the contrast to leave the pulmonary circulation, and enter the aorta and coronary arteries, a coronary CT angiography is performed within the same contrast bolus. No extra contrast is given to acquire the cardiac images. No intravenous beta-blocker nor sublingual nitroglycerin is administered.

The total added exam time (assessing heart rhythm, preparing the scan parameters, the delay time and the acquisition itself) is about one to two minutes.

The dose-length product (DLP) of the ECG-less cardiac scan depends on the duration of the scan time that is chosen. The average DLP is between 150 and 200 mGy.cm. The diagnostic reference level (DRL) as set by the Federal Agency for Nuclear Controle (FANC) for a coronary CT angiography is 300 mGy.cm.

The combined pulmonary CT angiography and ECG-less cardiac scan can be used to diagnose all the pathologies that can be assessed on a conventional pulmonary CT angiography scan (including, but not limited to, pneumonia, pleural fluid, pulmonary embolism, pulmonary infarct, pulmonary mass, pneumothorax, pericardial fluid, etc.) and provides extra diagnostic information about coronary artery disease.

In case the technique is well validated, future clinical questions could include whether ECG-less CCTA can help to identify a patient population of cardiac arrest survivors without STEMI that do benefit from early invasive coronary angiography and whether earlier treatment could improve outcome.

This study aims to investigate the feasibility and diagnostic accuracy of ECG-less gated CCTA in cardiac arrest survivors without STEMI, by means of agreement with ICA.

ELIGIBILITY:
* Inclusion:

  * Adults (≥18 years) with sustained return of spontaneous circulation (ROSC) following in/out-of-hospital cardiac arrest.
  * Informed consent from patient or representative obtained before invasive coronary angiography.
* Exclusion

  * Patients on VA-ECMO
  * ACS STEMI or STEMI "equivalent"

    * New left/right bundle branch block
    * ST segment depression in leads V1-V3, when the terminal T wave is positive and concomitant ST-segment elevation ≥ 0,5mm recorded in leads V7-V9 (posterior MI)
    * ST-segment elevation in V7-V9 (posterior MI) or V3R-V4R (RV MI)
  * ACS NSTEMI with persistent ST depression despite optimal therapy, suggesting ongoing myocardial ischemia, with indication for an urgent ICA according to the treating physician.
  * Hemodynamic/electrical instability precluding CT imaging (as perceived by the treating physician)
  * Life-threatening arrhythmia potentially caused by acute myocardial ischemia
  * Absolute contraindications to iodinated contrast
  * Patients with a known non-cardiac cause of cardiac arrest (e.g., traumatic brain injury, overt hemorrhage, asphyxia/severe hypoxia due to known lung disease, trauma, severe metabolic/electrolyte derangement, or intoxication) as perceived by the treating physician, where chest CT is considered unnecessary.
  * Known or likely pregnancy or lactation
  * Severe bleeding issue (as perceived by the treating physician) precluding heparin administration during radial access coronary angiography.
  * Prior coronary intervention (stent implantation/CABG).
  * CT findings indicating a condition that precludes coronary angiography in the short term.
  * Patients with end-of-life care pathways.
  * Participation in another intervention study interfering with the research questions in OPEN CCT Arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients correctly classified to coronary artery disease as the cause of cardiac arrest after analysis of the CT scan | Withing 24 hours after completion of the coronary angiography (which is performed within 24 hours of the CT scan) the comparative analysis will be performed
  With the invasive coronary angiography as a gold standard, the investigator will assess whether the CT scan correctly allocated the patient to coronary versus non coronary cause of cardiac arrest

SECONDARY OUTCOMES:
Level of agreement on the estimated percentage of coronary artery stenosis between CCTA and ICA | Withing 24 hours after completion of the coronary angiography (which is performed within 24 hours of the CT scan) the comparative analysis will be performed
  The degree of coronary stenosis will be estimated per-vessel (left main coronary artery, left anterior descendens, left circumflex artery and right coronary artery).
  The results will be reported as categorical variables: < 25%, 25-50%, 51-70%, 71-90%, >90% or insufficient image quality.
Feasibility of ECG-less gated CCTA in resuscitated patients | Within 24 hours after completion of the coronary angiography (which is performed within 24 hours of the CT scan) the analysis will be performed
  Percentage of patients where data on coronary stenosis based on ECG-less CCTA cannot be provided or is incompletely provided.
Reasons for failure of ECG-less gated CCTA image acquisition | Within 24 hours after completion of the coronary angiography (which is performed within 24 hours of the CT scan) the analysis will be performed
  Registrations of reasons for failure of complete CCTA reporting (eg incorrect timing, tachycardia/irregular heart rhythm...)
Survival | 90 days after enrollment
  Survival status assessed by analysis of the electronic medical record
Severe neurologic deficit | 90 days after enrollment
  Severe neurologic deficit definined as Modified Rankin Scale ≥ 3, assessed by consultation of the electronic health record (Y/N).
  The Modified Rankin Scale (mRS) is a scale used to assess the degree of disability or dependence. It is a 7-point scale, ranging from 0 (no symptoms) to 6 (death), designed to evaluate how well a patient can perform daily activities and how much assistance they need.
Peak troponin release | 90 days after enrollment
  Peak high sensitivity troponin T (ng/L) level during hospitalisation
Length of ICU stay | 90 days after enrollment
  Length of ICU stay (days)
Duration of catecholamine support | 90 days after enrollment
  Duration of catecholamine support (days) assessed by analysis of the electronic medical record
Peak SAPS II score | 90 days after enrollment
  The SAP II (Simplified Acute Physiology Score II) is a scoring system used to assess the severity of illness in critically ill patients, particularly those in intensive care units (ICU). It's designed to predict the risk of mortality based on various physiological variables measured in the first 24 hours of ICU admission.
  The score is calculated using 17 different clinical parameters, which include vital signs, lab results, and other physiological data. These parameters are categorized and assigned points, and the total score provides an estimate of the patient's risk of dying in the hospital.
  The score can range from 0 to 163. Higher scores indicate more severe illness and a higher risk of death.
Rehospitalization for heart failure | 90 days after enrollment
  Rehospitalization for heart failure (Y/N), assessed by analysis of the electronic medical record
Acute kidney injury (AKI) | 90 days after enrollment
  Development of AKI according to KDIGO definition (Y/N). AKI is diagnosed when there is a sudden decline in kidney function, defined by one of the following criteria:
  Serum Creatinine Criteria:
  * Stage 1: Increase in serum creatinine by ≥ 0.3 mg/dL (≥ 26.5 µmol/L) within 48 hours, or increase to 1.5-1.9 times baseline.
  * Stage 2: Increase in serum creatinine to 2.0-2.9 times baseline.
  * Stage 3: Increase in serum creatinine to 3.0 times baseline, or serum creatinine ≥ 4.0 mg/dL (≥ 354 µmol/L), or initiation of renal replacement therapy (dialysis), or in patients less than 18 years old, a decrease in glomerular filtration rate (GFR) to < 35 mL/min/1.73 m².
  Urine Output Criteria:
  Stage 1: Urine output < 0.5 mL/kg/hour for 6-12 hours. Stage 2: Urine output < 0.5 mL/kg/hour for ≥ 12 hours. Stage 3: Urine output < 0.3 mL/kg/hour for ≥ 24 hours, or anuria for ≥ 12 hours.
Need for renal replacement therapy (RRT) | 90 days after enrollment
  Need for renal replacement therapy (RRT) (Y/N)
ISTH major bleeding event | 90 days after enrollment
  Development of ISTH Major Bleeding Definition:
  According to the International Society on Thrombosis and Haemostasis (ISTH), a major bleeding event is one that involves at least one of the following:
  * Fatal Bleeding
  * Bleeding that Requires a Transfusion: requires the administration of 2 or more units of packed red blood cells (PRBCs) or equivalent blood products to treat blood loss.
  * Bleeding that Causes a Significant Drop in Hemoglobin: A decrease in hemoglobin of 2 g/dL or more or a hematocrit drop of ≥ 6%.
  * Bleeding that Requires Surgical Intervention
  * Intracranial Hemorrhage (ICH):
  * Other Severe Bleeding: Any other bleeding that is severe, for example, bleeding into a vital organ (e.g., bleeding into the eye causing loss of vision, or into the lungs causing respiratory compromise).
Ischemic stroke | 90 days after enrollment
  Development of ischemic stroke (Y/N)
Need for mechanical circulatory support (MCS) | 90 days after enrollment
  Need for mechanical circulatory support (MCS) (Y/N) Mechanical Circulatory Support (MCS) refers to the use of devices designed to support or assist the heart's ability to pump blood, typically in patients with acute or chronic heart failure. These devices are used to maintain or improve cardiac output in cases where the heart is not functioning adequately, often as a bridge to recovery, a bridge to heart transplantation, or as a long-term solution for patients who are not candidates for a transplant.
Treatment with Dual Antiplatelet Therapy (DAPT) | 90 days after enrollment
  Treatment with Dual Antiplatelet Therapy (DAPT) (Y/N)
LV systolic function | 90 days after enrollment
  Left ventricular systolic function assessed by ejection fraction (LVEF) on ambulatory follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel (UZB), Brussels, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Meier D, Andreini D, Cosyns B, Skalidis I, Storozhenko T, Mahendiran T, Assanelli E, Sonck J, Roosens B, Rotzinger DC, Qanadli SD, Tzimas G, Muller O, De Bruyne B, Collet C, Fournier S. Usefulness of FFR-CT to exclude haemodynamically significant lesions in high-risk NSTE-ACS. EuroIntervention. 2025 Jan 6;21(1):73-81. doi: 10.4244/EIJ-D-24-00779. PMID 39468963
- [Result] Meijboom WB, Meijs MF, Schuijf JD, Cramer MJ, Mollet NR, van Mieghem CA, Nieman K, van Werkhoven JM, Pundziute G, Weustink AC, de Vos AM, Pugliese F, Rensing B, Jukema JW, Bax JJ, Prokop M, Doevendans PA, Hunink MG, Krestin GP, de Feyter PJ. Diagnostic accuracy of 64-slice computed tomography coronary angiography: a prospective, multicenter, multivendor study. J Am Coll Cardiol. 2008 Dec 16;52(25):2135-44. doi: 10.1016/j.jacc.2008.08.058. PMID 19095130
- [Result] Budoff MJ, Dowe D, Jollis JG, Gitter M, Sutherland J, Halamert E, Scherer M, Bellinger R, Martin A, Benton R, Delago A, Min JK. Diagnostic performance of 64-multidetector row coronary computed tomographic angiography for evaluation of coronary artery stenosis in individuals without known coronary artery disease: results from the prospective multicenter ACCURACY (Assessment by Coronary Computed Tomographic Angiography of Individuals Undergoing Invasive Coronary Angiography) trial. J Am Coll Cardiol. 2008 Nov 18;52(21):1724-32. doi: 10.1016/j.jacc.2008.07.031. PMID 19007693
- [Result] Voicu S, Sideris G, Deye N, Dillinger JG, Logeart D, Broche C, Vivien B, Brun PY, Capan DD, Manzo-Silberman S, Megarbane B, Baud FJ, Henry P. Role of cardiac troponin in the diagnosis of acute myocardial infarction in comatose patients resuscitated from out-of-hospital cardiac arrest. Resuscitation. 2012 Apr;83(4):452-8. doi: 10.1016/j.resuscitation.2011.10.008. Epub 2011 Oct 29. PMID 22037386
- [Result] Staer-Jensen H, Nakstad ER, Fossum E, Mangschau A, Eritsland J, Draegni T, Jacobsen D, Sunde K, Andersen GO. Post-Resuscitation ECG for Selection of Patients for Immediate Coronary Angiography in Out-of-Hospital Cardiac Arrest. Circ Cardiovasc Interv. 2015 Oct;8(10):e002784. doi: 10.1161/CIRCINTERVENTIONS.115.002784. PMID 26453688
- [Result] Sideris G, Voicu S, Dillinger JG, Stratiev V, Logeart D, Broche C, Vivien B, Brun PY, Deye N, Capan D, Aout M, Megarbane B, Baud FJ, Henry P. Value of post-resuscitation electrocardiogram in the diagnosis of acute myocardial infarction in out-of-hospital cardiac arrest patients. Resuscitation. 2011 Sep;82(9):1148-53. doi: 10.1016/j.resuscitation.2011.04.023. Epub 2011 May 14. PMID 21632166
- [Result] Lee SE, Uhm JS, Kim JY, Pak HN, Lee MH, Joung B. Combined ECG, Echocardiographic, and Biomarker Criteria for Diagnosing Acute Myocardial Infarction in Out-of-Hospital Cardiac Arrest Patients. Yonsei Med J. 2015 Jul;56(4):887-94. doi: 10.3349/ymj.2015.56.4.887. PMID 26069108
- [Result] Dumas F, Manzo-Silberman S, Fichet J, Mami Z, Zuber B, Vivien B, Chenevier-Gobeaux C, Varenne O, Empana JP, Pene F, Spaulding C, Cariou A. Can early cardiac troponin I measurement help to predict recent coronary occlusion in out-of-hospital cardiac arrest survivors? Crit Care Med. 2012 Jun;40(6):1777-84. doi: 10.1097/CCM.0b013e3182474d5e. PMID 22488008
- [Result] Gonzalez MR, Esposito EC, Leary M, Gaieski DF, Kolansky DM, Chang G, Becker LB, Carr BG, Grossestreuer AV, Abella BS. Initial clinical predictors of significant coronary lesions after resuscitation from cardiac arrest. Ther Hypothermia Temp Manag. 2012 Jun;2(2):73-7. doi: 10.1089/ther.2012.0012. Epub 2012 Jul 9. PMID 24717160
- [Result] Desch S, Freund A, Akin I, Behnes M, Preusch MR, Zelniker TA, Skurk C, Landmesser U, Graf T, Eitel I, Fuernau G, Haake H, Nordbeck P, Hammer F, Felix SB, Hassager C, Engstrom T, Fichtlscherer S, Ledwoch J, Lenk K, Joner M, Steiner S, Liebetrau C, Voigt I, Zeymer U, Brand M, Schmitz R, Horstkotte J, Jacobshagen C, Poss J, Abdel-Wahab M, Lurz P, Jobs A, de Waha-Thiele S, Olbrich D, Sandig F, Konig IR, Brett S, Vens M, Klinge K, Thiele H; TOMAHAWK Investigators. Angiography after Out-of-Hospital Cardiac Arrest without ST-Segment Elevation. N Engl J Med. 2021 Dec 30;385(27):2544-2553. doi: 10.1056/NEJMoa2101909. Epub 2021 Aug 29. PMID 34459570
- [Result] Elfwen L, Lagedal R, Nordberg P, James S, Oldgren J, Bohm F, Lundgren P, Rylander C, van der Linden J, Hollenberg J, Erlinge D, Cronberg T, Jensen U, Friberg H, Lilja G, Larsson IM, Wallin E, Rubertsson S, Svensson L. Direct or subacute coronary angiography in out-of-hospital cardiac arrest (DISCO)-An initial pilot-study of a randomized clinical trial. Resuscitation. 2019 Jun;139:253-261. doi: 10.1016/j.resuscitation.2019.04.027. Epub 2019 Apr 24. PMID 31028826
- [Result] Thevathasan T, Freund A, Spoormans E, Lemkes J, Rossberg M, Skurk C, Fichtlscherer S, Akin I, Fuernau G, Hassager C, Zeymer U, Preusch MR, Graf T, Jung C, Abdel-Wahab M, Jobs A, Laufs U, Schulze PC, Linke A, de Waha S, Poss J, Thiele H, Desch S. Bayesian Reanalyses of the Trials TOMAHAWK and COACT. JACC Cardiovasc Interv. 2024 Dec 23;17(24):2879-2889. doi: 10.1016/j.jcin.2024.09.071. PMID 39722271
- [Result] Lemkes JS, Janssens GN, van der Hoeven NW, Jewbali LSD, Dubois EA, Meuwissen M, Rijpstra TA, Bosker HA, Blans MJ, Bleeker GB, Baak R, Vlachojannis GJ, Eikemans BJW, van der Harst P, van der Horst ICC, Voskuil M, van der Heijden JJ, Beishuizen A, Stoel M, Camaro C, van der Hoeven H, Henriques JP, Vlaar APJ, Vink MA, van den Bogaard B, Heestermans TACM, de Ruijter W, Delnoij TSR, Crijns HJGM, Jessurun GAJ, Oemrawsingh PV, Gosselink MTM, Plomp K, Magro M, Elbers PWG, van de Ven PM, Oudemans-van Straaten HM, van Royen N. Coronary Angiography after Cardiac Arrest without ST-Segment Elevation. N Engl J Med. 2019 Apr 11;380(15):1397-1407. doi: 10.1056/NEJMoa1816897. Epub 2019 Mar 18. PMID 30883057
- [Result] ESC Scientific Document Group. [2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death]. G Ital Cardiol (Rome). 2023;24(3 Suppl 1):e1-e132. doi: 10.1714/3986.39669. No abstract available. Italian. PMID 36880552

DOCUMENTS (2):
  • Study Protocol (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT07388342/Prot_000.pdf
  • Informed Consent Form (2025-06-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT07388342/ICF_001.pdf